CLINICAL TRIAL: NCT01487928
Title: A Randomized Study of the Use of Human Milk Cream as a Caloric Supplement in a Subset of Very Low Birth Weight Pre-Term Infants
Brief Title: Human Milk Cream as a Caloric Supplement in Pre-Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Prolacta Bioscience (Industry)
Responsible Party: Principal Investigator, Amy Hair, Assistant Professor of Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-29743
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prematurity
Keywords: breastfed; human milk cream; human milk fat; caloric supplement
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Human Milk Cream Group (Experimental): For infants randomized to the human milk cream group, the human milk (either mother's own or donor) being provided to the infant will be tested each time a new container is used to prepare feedings. The test will be for the caloric content of the milk using a commercially available device provided for this purpose. If the caloric level falls below 20 kcal/oz for any test, then an appropriate amount of human milk cream will be added to the milk to bring the content as close as possible to 20 kcal/oz. The amount added will be calculated to the nearest mL rounding down for 0.1-0.4mL and up for 0.5-0.9 mL to avoid imprecision due to the measuring device used in the nutrition preparation area.
  Interventions: Dietary Supplement: Human Milk Cream
- Control Group (No Intervention): For infants randomized to the Control group, human milk and human milk derived fortifier will be provided according to the institutional standard of care and there will be no use of the milk analysis (mother's own or donor), which is typical for the vast majority of neonatal intensive care units.

INTERVENTIONS:
Dietary Supplement: Human Milk Cream — If the caloric level of human milk (mother's own or donor) falls below 20 kcal/oz, then an appropriate amount of human milk cream will be added to the milk to bring the content as close as possible to 20 kcal/oz. For example, if the human milk is 19 kcal/oz, 2 mL of human milk cream will be added to 100mL of human milk.
  Arms: Human Milk Cream Group

SUMMARY:
Human milk is commonly considered to have 20 calories per ounce (kcal/oz). However, studies show that up to 65% of human milk may be less than the expected 20 kcal/oz which can greatly affect an infant's growth. The investigators now have the ability to measure caloric density of human milk and add human milk cream to any human milk (mother's own or donor human milk) that is less than 20 kcal/oz to bring it up to that amount.

DETAILED DESCRIPTION:
Once fortification (to either mother's or donor milk) is initiated and tolerance is established (based on clinical observation), infants will be randomized into one of two groups: to receive human milk cream or not.

* Human Milk Cream Group: Human milk (either mother's own or donor) will be tested (once per container of milk). If the caloric level falls below 20 kcal/oz, then an appropriate amount of human milk cream will be added to the milk to bring the content as close as possible to 20 kcal/oz.
* Control Group (no human milk cream): Milk (either mother's own or donor) and human milk fortifier will be provided as usual (milk will be analyzed for study purposes).

This nutritional algorithm will continue until the infant reaches 36 weeks corrected gestational age/weaned from fortifier (whichever comes first) or is otherwise removed from the study (due to transfer to non-study institution, removal from the study or death).

Data will be collected from the time of study entry until the infant reaches 36 weeks corrected gestational age or weaned from the fortifier (whichever comes first) or is otherwise removed from the study.

Primary measure of efficacy:

The primary measure of efficacy for the study is the rate of change of weight from the initiation of enteral feeding through 36 weeks corrected gestational age or weaned from fortifier, whichever comes first. Based on an intent-to-treat (ITT) paradigm, if a study subject fails to complete the study period for any reason, this rate will be determined for the period of time on study. In order to provide a valid comparison between the study subjects, the rate of weight gain will be reported as g/kg/day. In a per-protocol analysis, these subjects will be dropped from any calculations with respect to this primary endpoint.

Primary measure of safety:

For the evaluation of safety, any untoward effects deemed to be related to the nutritional regimen will be identified and recorded. Key outcomes in this regard include feeding intolerance, necrotizing enterocolitis (NEC) and sepsis. Because this population has a high associated morbidity, episodes of apnea, and the use of oxygen and ventilators will be evaluated from a safety perspective.

Baseline measures: (study entry, i.e. initiation of enteral feeding)

At study entry, the following variables will be recorded: birth weight, gestational age, gender, Apgar score at 5 minutes, use of mechanical ventilation at study entry, use of prenatal or postnatal steroids, and the age in days at which enteral feeding was initiated. In addition the presence of any of the following clinical conditions either at the time of study entry or occurring during the course of the study will be noted: transient tachypnea of newborn (TTN), intraventricular hemorrhage (IVH) and grade, and patent ductus arteriosis (PDA).

Other growth measures:

Head circumference increment for the study period and length increment for the study period will be determined (and recorded as cm/week). Length and head circumference will be recorded on a weekly basis during the study period. The use of medications that influence growth and development will be recorded. These include postnatal steroids, e.g. hydrocortisone and dexamethasone, caffeine and other methylxanthine preparations.

Feeding protocol:

The daily amount of all enteral nutrition will be recorded in units of mL. This quantity will be subdivided into the various types of nutrition used, i.e. mother's milk, donor milk, human milk cream, fortifiers, and any other nutritional support. In the event of feeding intolerance or discontinuation of enteral feeding and the baby being returned to total parenteral nutrition (TPN), the assumed cause will be identified. The total number of days of TPN will be recorded for the study period as well as the range of dates the infant was on TPN.

Infectious complications:

Although not a focus of this study, occurrences of sepsis, NEC and other related infectious outcomes will be recorded.

Demographics:

Basic demographic and medical information on each subject will be collected and recorded. These variables include: gestational age, birth weight (including whether the infant was AGA or SGA based on standard criteria), gender, and racial group.

Medications:

Information on the dosing of the following drugs will be recorded: Lasix, caffeine, diuril, insulin, and dopamine.

Parenteral Nutrition:

Components and rate of parenteral nutrition will be recorded during study days to further evaluate nutritional intake and growth.

Labs:

Nutritionally-relevant labs that are obtained for clinical purposes will be recorded: Na, K, Cl, CO2, BUN, Creatinine, glucose, Ca, Phos, Mg, and triglycerides.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight 750 - 1250g
* Able to adhere to expected feeding protocol of mother's own milk/donor milk with fortification of Prolacta® fortifier
* Reasonable expectation of survival
* Enteral feeding must begin before the 21st day of life

Exclusion Criteria:

* Decision to not start minimum enteral feed before day 21 of life
* Unable to obtain informed consent from parent/guardian prior to the initiation of fortification of enteral feeding
* Enrolled in any other clinical study affecting nutritional management during the study period
* Presence of clinically significant congenital heart disease or major congenital malformations
* Reasonable potential for early transfer to a non-study institution

Max Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2011-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Caloric content of human milk | Daily until 36 weeks corrected gestational age
  Human milk samples will be analyzed for macronutrients and total caloric content.

SECONDARY OUTCOMES:
Growth | Weekly until 36 weeks corrected age
  Growth (weight, length, and head circumference) will be evaluated weekly throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Amy B Hair, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor College of Medicine / Texas Children's Hospital, Houston, Texas
  - UT Health Science Center, San Antonio, San Antonio, Texas

REFERENCES:
- [Background] Sullivan S, Schanler RJ, Kim JH, Patel AL, Trawoger R, Kiechl-Kohlendorfer U, Chan GM, Blanco CL, Abrams S, Cotten CM, Laroia N, Ehrenkranz RA, Dudell G, Cristofalo EA, Meier P, Lee ML, Rechtman DJ, Lucas A. An exclusively human milk-based diet is associated with a lower rate of necrotizing enterocolitis than a diet of human milk and bovine milk-based products. J Pediatr. 2010 Apr;156(4):562-7.e1. doi: 10.1016/j.jpeds.2009.10.040. Epub 2009 Dec 29. PMID 20036378
- [Background] Wojcik KY, Rechtman DJ, Lee ML, Montoya A, Medo ET. Macronutrient analysis of a nationwide sample of donor breast milk. J Am Diet Assoc. 2009 Jan;109(1):137-40. doi: 10.1016/j.jada.2008.10.008. PMID 19103335
- [Background] Hawthorne KM, Griffin IJ, Abrams SA. Current issues in nutritional management of very low birth weight infants. Minerva Pediatr. 2004 Aug;56(4):359-72. PMID 15457134
- [Derived] Fabrizio V, Trzaski JM, Brownell EA, Esposito P, Lainwala S, Lussier MM, Hagadorn JI. Individualized versus standard diet fortification for growth and development in preterm infants receiving human milk. Cochrane Database Syst Rev. 2020 Nov 23;11(11):CD013465. doi: 10.1002/14651858.CD013465.pub2. PMID 33226632
- [Derived] Amissah EA, Brown J, Harding JE. Protein supplementation of human milk for promoting growth in preterm infants. Cochrane Database Syst Rev. 2020 Sep 23;9(9):CD000433. doi: 10.1002/14651858.CD000433.pub3. PMID 32964431
- [Derived] Hair AB, Blanco CL, Moreira AG, Hawthorne KM, Lee ML, Rechtman DJ, Abrams SA. Randomized trial of human milk cream as a supplement to standard fortification of an exclusive human milk-based diet in infants 750-1250 g birth weight. J Pediatr. 2014 Nov;165(5):915-20. doi: 10.1016/j.jpeds.2014.07.005. Epub 2014 Aug 15. PMID 25130571